CLINICAL TRIAL: NCT03240055
Title: The Effects of Spinal Anesthesia on ED50 and BIS50 of Etomidate for the Loss of Consciousness
Acronym: LOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: mz2017
Record Dates: First submitted 2017-07-21; First posted 2017-08-04 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Dose-Response Relationship, Drug
Keywords: spinal anesthesia; etomidate; median effective dose; BIS50
MeSH Terms: interventions — Anesthesia, Spinal; Etomidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SE (Experimental): 21 patients received spinal anesthesia first. After confirmation of the level (T4-T6) of the sensory anesthesia, the sequential administration of etomidate was conducted
  Interventions: Drug: spinal anesthesia
- Group E (Placebo Comparator): 27 patients without spinal anesthesia in this group received sequential administration of etomidate
  Interventions: Other: etomidate

INTERVENTIONS:
Drug: spinal anesthesia — The spinal puncture was performed with a 25 G Sprotte needle at the L3-4 or L2-3 interspinous space. Hyperbaric bupivacaine 0.5% (3 ml) was administered into the spinal space. Hyperbaric bupivacaine is obtained through the addition of glucose 10% (1ml) to bupivacaine 0.75% (2ml). Cerebrospinal fluid aspiration (0.1 ml) was done to confirm correct needle placement before and after spinal drug administration. Whereafter the patient was turned rapidly to the supine position, sensory anesthesia height was evaluated bilaterally using a pinprick test with the sharp tip of a safety pin every 1 min until 15 min after the initiation of the spinal anesthesia, bed tilting (upwards, horizontal, or downwards) was performed until bilateral sensory anesthesia level was confirmed to remain at the T4-T6 level
  Arms: Group SE
Other: etomidate — receive etomidate only
  Arms: Group E

SUMMARY:
The purpose of this study is to investigate the effect of spinal anesthesia on ED50 and BIS50 of etomidate for the loss of consciousness (LOC) by using up-and-down method.The hypothesis was that spinal anesthesia could significantly reduce the etomidate bolus dose for the LOC and could also achieve hemodynamic stability during anesthesia induction.

DETAILED DESCRIPTION:
The combination of spinal with general anesthesia has been demonstrated to provide many clinically relevant advantages, however, this technique often experiences hypotension and bradycardia in the induction period of combined anesthesia. Etomidate is a carboxylated imidazole-derived hypnotic, and it is the most cardiovascularly stable intravenous induction drug, with the possible exception of ketamine. Meanwhile, the previous and our studies have been reported that spinal anesthesia has a direct sedative effect on animals and humans, and it markedly reduces the dose of hypnotic agents. To date, there is no dose-ranging study on the effect of spinal anesthesia on dosage of etomidate for the loss of consciousness (LOC). In the present study, investigators aim to investigate the effect of spinal anesthesia on the median effective dose (ED50) and the BIS value (BIS50) of etomidate at which 50% of patients lose consciousness compared to etomidate alone by using up-and-down method.

Patients were randomly allocated to one of two groups: only etomidate in group E (n=27) and spinal anesthesia combined with etomidate in group SE (n=21) using a randomization table. Patients in the SE group received spinal anesthesia first, and bilateral sensory anesthesia level was confirmed to remain at the T4-T6 level. After confirmation of the level of sensory anesthesia, the administration of etomidate was conducted. The etomidate (Nhwa Pharmaceutical, Jiangsu, China) starting dose of E group and SE group is 0.105 mg/kg and 0.089mg/kg, respectively. The dose of etomidate used for next patient was determined according to the response of the previously tested patient using the up-and-down method. If the patient lose consciousness, the dose of etomidate was reduced by one dose gradient for the next patient, and if didn't lose consciousness, the dose of etomidate was increased by one dose gradient (one dose gradient is r=1:0.85, that is, the ratio of high dose/low dose which are adjacent two doses). The testing of different dose levels of etomidate continued on consecutive randomised patients until a sample size of seven crossover points from "conscious" to "LOC" was reached

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Body mass index (BMI) between 18.0 and 24.5 kg/m2
* Undergoing short elective laparotomy procedures, hysteroscopic and vaginal operation

Exclusion Criteria:

* Contraindication to spinal anesthesia
* Hearing loss
* History of cardiovascular disease, psychiatric and central nervous system diseases
* Hepatic or renal dysfunction
* Severe diabetes or hyperkalemia
* History of drug and alcohol abuse
* An allergy to amide local anesthetics or etomidate
* Adrenocortical hypofunction

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Median effective dose (ED50)of etomidate at which 50% of patients lose consciousness | After etomidate administration to the lowest BIS value appears，usually about 4 minutes
  We want to determine Median effective dose (ED50) of etomidate at which 50% of patients lose consciousness in the SE and E group, respectively. It is a value，like 0.105mg/kg. Patients were considered to be loss of consciousness if there Observer's Assessment of Alertness/Sedation (OAA/S) scores were 2,1,or 0.
BIS value (BIS50) of etomidate at which 50% of patients lose consciousness | After etomidate administration to the lowest BIS value appears，usually about 4 minutes
  We want to determine BIS value (BIS50) of etomidate at which 50% of patients lose consciousness in the SE and E group, respectively. It is a unitless value，like 60. Patients were considered to be loss of consciousness if there Observer's Assessment of Alertness/Sedation (OAA/S) scores were 2,1,or 0.

SECONDARY OUTCOMES:
The change of Mean Arterial Pressure (MAP) | Baseline, l min (T1), 2min (T2), 3min (T3), 5min (T5) after administration of etomidate
The change of heart rate (HR) | Baseline, l min (T1), 2min (T2), 3min (T3), 5min (T5) after administration of etomidate

CONTACTS AND LOCATIONS:
Overall Officials: Li Ningkang, Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No
safety